CLINICAL TRIAL: NCT04331340
Title: A Project to Address Lower Urinary Tract Symptoms (LUTS) by Pharmacists in the Community
Brief Title: Management of LUTS by Community Pharmacists
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00097144
Record Dates: First submitted 2020-03-23; First posted 2020-04-02 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Lower Urinary Tract Symptoms
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacist Intervention (Experimental): Pharmacist assessment of LUTS, with recommendations and education regarding lifestyle, behaviour, and/or medications related to bladder health. Follow-up at 3 and 6 weeks.
  Interventions: Other: Pharmacist review of LUTS
- Control (Active Comparator): Pharmacist questions regarding presence of LUTS, with provision of healthy aging literature. Follow-up at 6 weeks.
  Interventions: Other: Pharmacist Provision of healthy aging leaflets

INTERVENTIONS:
Other: Pharmacist review of LUTS — Pharmacist review and recommendations, including education, behaviour, lifestyle, or medications
  Arms: Pharmacist Intervention
Other: Pharmacist Provision of healthy aging leaflets — Pharmacist will inquire about presence of LUTS and provide patient with healthy aging leaflets
  Arms: Control

SUMMARY:
Many older adults have urinary incontinence. They often seek treatments, such as diapers, pads, or medications, from the community pharmacy. Pharmacists are trained to assist seniors with therapies that treat urinary incontinence. Our study will determine how much benefit there is if pharmacists try to provide more assistance for seniors with incontinence. Over a period of months, half of the people who talk to the pharmacist about their incontinence will be given general information about health and aging. The other half of the people will have a longer assessment and complete a questionnaire with the pharmacist. Then the pharmacist will call and have a follow-up visit to see how the incontinence symptoms have improved. We will compare both groups to see whose symptoms were improved.

DETAILED DESCRIPTION:
This randomized controlled trial is designed to determine the effect of a pharmacist intervention to manage lower urinary tract symptoms (LUTS) in the community. The objectives of the study are to determine the effect of the pharmacist as measured by the Patient Perception of Bladder Condition (PPBC) (primary objective), the Bladder Self-Assessment Questionnaire (B-SAQ), and the International Consultation on Incontinence Module Questionnaire Short Form (ICI-Q-SF) (as secondary objectives).

The pharmacists at community pharmacies will be recruited through the networks already established within Alberta for pharmacy practice research, and the Pharmacists Association of Alberta. The pharmacists must have advanced prescribing authorization with their professional license.

The patients will be recruited with the posting of shelf-talkers by the incontinence and menstrual products section of the pharmacy and with leaflets in prescription bags. If a patient obtains a LUTS product or if the patient presents him/herself in response to the shelf-talker, the pharmacist will screen the patient to determine if LUTS are present.The patients will be eligible to participate if they are at least 60 years of age, report LUTS, can communicate in English, and provide consent.

The patient will be randomized to either a control or intervention. Those assigned to the control group will be eligible to receive the intervention following the follow-up period. Both the control and intervention group will have a baseline PPBC, B-SAQ, and ICI-Q-SF questionnaires, in addition to demographics and a medical history.

The control group will receive a healthy aging pamphlet and will be called back at 8 weeks to have the questionnaires repeated.

The intervention is based on the published guide for LUTS for pharmacists (Gabriel, et al. 2015). The pharmacist will assess the patient's LUTS and determine an appropriate intervention plan, which may include education, lifestyle, behavioural, or medication modification. The patient will be given a summary of the plan and the primary care provider will also receive a summary. At 4 weeks the patient will be contacted by phone or in person (per patient preference), with a review of the plan and repeated bladder questionnaires. At 8 weeks the patient will complete the final interaction with the pharmacist and will complete the bladder questionnaires for the final time.

The primary outcome is the change in PPBC from baseline to 8 weeks, and secondary outcomes include the change from baseline until 8 weeks in the B-SAQ, ICI-Q, and health system use (including referrals to physicians, specialists, and pharmacist billing).

We plan to enroll 100 patients (50 in each group). All analyses will be by intention to treat.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥60 years
* Report lower urinary tract symptoms (LUTS)
* Read and communicate in English

Exclusion Criteria:

* Age ≤ 59 years
* Deny LUTS
* Refuse to consent
* Unavailable or unable to participate in follow-up visits

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Patient Perception of Bladder Condition (PPBC) | Change from baseline to 8 weeks post-intervention
  Questionnaire to assess patient perception of LUTS severity Scored from 1-6; 1 = problems, 6=severe problems

SECONDARY OUTCOMES:
Change in Bladder Self-Assessment Questionnaire (B-SAQ) | Change from baseline to 8 weeks post-intervention
  Self-administered questionnaire to assess types of symptoms and extent of bother Scored for Bother 0-12; 0=no bother, 12 = bothers a great deal Scored for Symptoms 0-12; 0=no symptoms, 3=severe symptoms
Change in International Consultation on Incontinence Module Questionnaire Short Form (ICI-Q-SF) | Change from baseline to 8 weeks post-intervention
  Self- administered questionnaire to describe extent and severity of LUTS Scored from 0-21; 0= no impact or leakage; 21 = severe leakage and interference

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl A Sadowski, Pharm.D., Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
Subject demographics and scores of the primary and secondary outcomes measures will be shared at all time points.
Time Frame: After completion of the study in 2021, for 5 years.